CLINICAL TRIAL: NCT04292054
Title: "Antibioprophylaxis for Excision-graft Surgery in Burn Patient: a Multicenter Randomized Double-blind Study: A2B Trial"
Brief Title: Antibioprophylaxis for Excision-graft Surgery in Burn Patient (A2B-TRIAL)
Acronym: A2B
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP180605
Record Dates: First submitted 2020-02-17; First posted 2020-03-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Burns Surgery
Keywords: Antibioprophylaxis; sepsis; infection; graft lysis
MeSH Terms: conditions — Sepsis; Infections | interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled study with two arms (1:1)
  Arm 1 : With antibiotic prophylaxis strategy, (cefazolin) if absence of colonization to Pseudomonas aeruginosa; or (piperacilline-tazobactam) if the burn is colonized with Pseudomonas aeruginosa.
  Arm 2 : Without antibiotic prophylaxis strategy (placebo)
Who Masked: Participant, Investigator
Masking Description: Treatments will be conditioned by the Contract manufacturing organization (central pharmacy of Assistance-Publique Hôpitaux de Paris) according to a list provided by an independent person and assigning a treatment arm to each treatment number
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active group (Active Comparator): The antibiotic prophylaxis will be cefazolin 2 g powder for solution for injection diluted in 50mL of NaCl 0.9%, IV infusion on 30 minutes with syringe pump, in case of absence of colonization to Pseudomonas aeruginosa prior to the surgical procedure.
  The dose administer is 2g.
  Antibiotic prophylaxis will be piperacilline-tazobactam 4 g powder for solution for injection diluted in 50mL of NaCl 0.9%, IV infusion on 30 minutes with syringe driver in patients with burn wound colonized to Pseudomonas aeruginosa.
  The dose administer is 4g.
  Interventions: Drug: active intervention
- Placebo group (Placebo Comparator): The control group will received, as placebo NaCl 0.9% solution for injection diluted in 50mL of NaCl 0.9%, IV infusion on 30 minutes with syringe pump.
  Interventions: Other: placebo intervention

INTERVENTIONS:
Drug: active intervention — The antibiotic prophylaxis will be cefazolin 2 g, or piperacilline-tazobactam 4 g, powder for solution for injection diluted in 50mL of NaCl 0.9%, IV infusion on 30 minutes with syringe pump.
  Other Names: Cefazolin or piperacilline-tazobactam 4 g
  Arms: active group
Other: placebo intervention — The control group will received, as placebo NaCl 0.9% solution for injection diluted in 50mL of NaCl 0.9%, IV infusion on 30 minutes with syringe pump.
  Other Names: NaC 0,9%l
  Arms: Placebo group

SUMMARY:
The indication of antibiotic prophylaxis in burn patients remains highly controversial and hasn't reached a consensus. The objective of antibiotic prophylaxis would be to reduce the risk of post-operative local and systemic infections. Burn surgery is associated with a high risk of bacteremia and postoperative infections and sepsis. However, antibiotic prophylaxis exposes to the risk of selecting drug-resistant pathogens as well as adverse effects of antibiotics (i.e Clostridium difficile colitis).

Recommendations regarding perioperative prophylaxis using systemic antibiotics vary across sources. The lack of data precludes any international strong recommendations regarding the best strategy regarding antibiotic prophylaxis.

The goal of this project is therefore to determine whether peri-operative systemic antibiotics prophylaxis could reduce the incidence of post-operative infections in burn patients.

DETAILED DESCRIPTION:
The intensive care unit investigator will verify the inclusion and non-inclusion criteria.

The following parameters will be collected at ICU/burn centers: Hemodynamic parameters; sepsis organ failure assessment (SOFA) score, Glasgow Coma scale; Medical history / comorbidities; Concomitant treatment; Burn wound bacterial colonization; Biological parameters.

The inclusion and randomization will be performed as late as possible before the first surgical procedure.

Randomization: Burn patients with deep burn between 5 to 40% TBSA requiring at least one excision surgery graft will be randomized to receive antibioprophylaxis (or placebo) 30 minutes before the incision with either first generation cephalosporin (cefazolin) (if absence of colonization to Pseudomonas aeruginosa); or piperacillin-tazobactam (if the burned area is colonized with Pseudomonas aeruginosa). We chose to target specifically Pseudomonas aeruginosa because it has been associated with significant morbidity and risk of graft lysis in burn patients.

No specific exams are required during the 7 days, 28 days and 90 days follow up visits.

The end of research visit is the 90-day follow-up visit. If the patient has been discharged from the hospital, the 90-day visit will consist of a telephone contact with the patient if he or she has been discharged home or with the medical team of the healthcare structure if the patient has been discharged to another structure.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years and less than 80 years old
* Burned patients requiring at least one excision-graft surgery
* Burn TBSA% between 5% and 40%
* Signed informed consent or inclusion under the emergency provisions of the law (article L1122-1-2 of the CSP)

Exclusion Criteria:

* Proven severe allergy to cephalosporin or piperacilline-tazobactam or any other antibacterial agent of the penicillin class
* History of severe allergic reaction to any other beta-lactam (eg cephalosporins, monobactams or carbapenems).
* Patient on antibiotic therapy at the time of surgery
* Pregnant or breast-feeding patient
* Patient not covered by the social security
* Patient transferred from another burn Unit
* Patient participant in investigational competitive medicinal product study on the primary endpoint
* Patient with local or systemic signs of infection requiring systemic antimicrobial therapy
* Patient under guardianship
* Patient under curatorship
* known colonization of the burned area to be excised with tazocillin-resistant germ.
* obese patient with BMI > 50 kg/m²

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative infection defined as Post-operative sepsis and/or Surgical site infection, and/or Graft lysis requiring a new graft within 7 days after surgery. | 7 days after surgery
  Postoperative infection will be collected by the intensivists or infectious disease specialist consultant blinded to the interventional or control arm. Skin infection and skin graft lysis requiring a new graft procedure will be assess by a surgeon blinded of the arm of the study.
Post-operative sepsis | 7 days after surgery
  Sepsis is defined as life-threatening organ dysfunction (defined by an increase of Sepsis related organ failure assessment [SOFA] score of 2 points or more) in response to infection. The minimum value is 0 and maximum value is 24. 0 meaning no organ dysfunction and 24 the maximum organ dysfunction.
Surgical site infection | 7 days after surgery
  Surgical site (operated skin) infection with general signs is considered as a systemic infection originated from skin (Presence of a local or loco-regional inflammatory reaction; Unfavourable and unexpected local evolution; Lysis of grafts; Necrosis of fat located under the graft)
Graft lysis needing a new graft procedure | 7 days after surgery
  Graft lysis is defined as a skin graft lysis in the 7 days post operative, and needing a new skin graft assessed be a surgeon blinded of the randomization group.

SECONDARY OUTCOMES:
Mortality | At day 90
  Any death occurring between randomization and D 90
Skin graft lysis requiring a new graft procedure | 7 days after surgery
  Defined as a skin graft lysis in the 7 days post operative, and needing a new skin graft assessed be a surgeon blinded of the randomization group.
Postoperative bacteremia | within 7 days of surgery
  Positive blood culture .
Post-operative pulmonary infection | 7 days after surgery
  Imaging Test Evidence
  Two or more serial chest imaging test results with at least one of the following:
  New and persistent or Progressive and persistent
  * Infiltrate
  * Consolidation
  * Cavitation Signs/Symptoms/Laboratory
  For ANY PATIENT, at least one of the following:
  * Fever (>38.0°C or >100.4°F)
  * Leukopenia (≤4000 WBC/mm) or leukocytosis (>12,000 WBC/mm)
  * For adults >70 years old, altered mental status with no other recognized cause
  And at least two of the following:
  * New onset of purulent sputum or change in character of sputum, or increased respiratory secretions, or increased suctioning requirements
  * New onset or worsening cough, or dyspnea, or tachypnea
  * Rales or bronchial breath sounds
  * Worsening gas exchange
Post-operative surgical site infection | 7 days after surgery
  Skin infection with general signs is considered as a systemic infection originated from skin.
Number of hospitalization days living without antibiotic therapy | at Day 28 and Day 90
  It will be calculated as the number of survival days without antibiotic therapy respectively between randomization and day 28 and day 90.
Number of days of hospitalization until complete healing (> 95% total burn surface area) | at Day 28 and Day 90
  It will be calculated by the number of days between ICU complete healing and ICU discharge.
Number of patients with a colonization with a multidrug resistant bacteria. | at Day 28 and Day 90
  It will be defined as :
  AmpC producer enterobacteriacae Extended spectrum beta lactamase enterobacteriacae Carbapenemase producer enterobacteriacae Meticillin resistant aureus staphylococcus Vancomycine resistant enterococcus Piperacillin-Tazobactam resistant bacteria Imipenem resistant Acinetobacter Baumanii. And it will be mesured from results of bacterial cultures and/or genotyping with antibiogramm resistance profile

CONTACTS AND LOCATIONS:
Overall Officials: François DEPRET, MD, Principal Investigator — Department of Anesthesiology, Critical Care and Burn Unit; Saint-Louis hospital
Locations (1):
- Saint Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Depret F, Farny B, Jeanne M, Klouche K, Leclerc T, Nouette-Gaulain K, Pantet O, Remerand F, Roquilly A, Rousseau AF, Sztajnic S, Wiramus S, Vicaut E, Legrand M; A2B trial investigators. The A2B trial, antibiotic prophylaxis for excision-graft surgery in burn patients: a multicenter randomized double-blind study. Trials. 2020 Nov 25;21(1):973. doi: 10.1186/s13063-020-04894-y. PMID 33239101